CLINICAL TRIAL: NCT03338127
Title: Outcomes of Acute Kidney Injury in Critically Ill Patients in Luxor International Hospital
Brief Title: Outcomes of Acute Kidney Injury in Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Alaa H Fahmy (Other)
Responsible Party: Sponsor-Investigator, Alaa H Fahmy, Principal Investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: AssiutU AHFahmy
Record Dates: First submitted 2017-11-01; First posted 2017-11-09 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Kidney Function Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: all patients recruited in the trial will be investigated for renal function test
  Interventions: Diagnostic Test: renal function test

INTERVENTIONS:
Diagnostic Test: renal function test — 2 ml blood sample to be investigated for renal function test

SUMMARY:
this study to evaluate the frequency of acute kidney injury in critically ill patients in intensive care units.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) affects approximately 20% of hospitalized patients and up to 67% of those admitted to an intensive care unit (ICU), making it among the most common organ dysfunctions among the critically ill . Depending on severity, Acute kidney injury (AKI) contributes to short-perimortality rates between 40% and 70% , and survivors are at increased risk for chronic kidney disease (CKD) and late death.

The diagnosis of Acute kidney injury (AKI) is only considered after achieving an adequate status of hydration and after excluding urinary obstruction; Acute kidney injury (AKI) is defined by the sudden decrease (in 48 h) of renal function, defined by an increase in absolute serum creatinine of at least (0.3 mg/dL) or by a percentage increase in serum creatinine ≥50% (1.5× baseline value), or by a decrease in the urinary output (documented oliguria <0.5 mL/kg/h for more than 6hours).

The purpose of this study was to benchmark the outcomes of acute kidney injury in a critically ill surgical patients.We hypothesized that renal dysfunction in this population is common and is associated with a significantly higher burden of morbidity, mortality, and resource utilization

ELIGIBILITY:
Inclusion Criteria:

• All patient with acute kidney injury in critical care units in Luxor international hospital

Exclusion Criteria:

* Patients on chronic dialysis
* Previous acute kidney injury
* Nephrectomy
* Organ transplant
* Chronic kidney disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient willl be recruited from critical care units in Luxor international hospital
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury in critically ill patients | 10 days
  To evaluate the frequency of acute kidney injury in critically ill patients admitted in intensive care units.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Aly, professor, Study Director — professor of internal medicine

IPD SHARING:
Plan to Share IPD: Undecided